CLINICAL TRIAL: NCT05292586
Title: A 12 Week, Randomized, Double-blind, Multicenter, Active Controlled, 2-Arm Parallel Group Study Testing the Superiority of CHF 1535 pMDI 800/24µg Total Daily Dose (Fixed Combination of Extrafine Beclomethasone Dipropionate Plus Formoterol Fumarate) Compared to CHF 718 pMDI 800µg Total Daily Dose (Extrafine Beclomethasone Dipropionate) in Adults With Asthma on Medium or High-Dose Inhaled Corticosteroid
Brief Title: A Study Testing the Superiority of CHF 1535 pMDI 800/24µg Total Daily Dose Compared With CHF 718 pMDI 800µg Total Daily Dose in Adults With Asthma on Medium or High-Dose Inhaled Corticosteroid
Acronym: FORCE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-05993AB8-02
Record Dates: First submitted 2022-03-04; First posted 2022-03-23 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Asthma
Keywords: Asthma; Beclomethasone Dipropionate; Beclometasone dipropionate/Formoterol fumarate; Inhaled Corticosteroids; CHF 1535 pMDI; CHF 718 pMDI
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinded roles were participant, investigator, care provider, monitor, data analyst, and assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CHF 1535 pMDI (Experimental): CHF 1535 pMDI 800/24µg TDD
  Interventions: Drug: Beclomethasone Dipropionate/Formoterol Fumarate
- CHF 718 pMDI (Active Comparator): CHF 718 pMDI 800µg TDD
  Interventions: Drug: Beclomethasone Dipropionate

INTERVENTIONS:
Drug: Beclomethasone Dipropionate/Formoterol Fumarate — Available in pressurized inhalation solution BDP/FF 200/6 µg
  Other Names: BDP/FF
  Arms: CHF 1535 pMDI
Drug: Beclomethasone Dipropionate — Available in pressurized inhalation solution BDP 100 µg
  Other Names: BDP
  Arms: CHF 718 pMDI

SUMMARY:
Compare the superiority of CHF 1535 versus CHF 718 in subjects with asthma who are on medium or high dose inhaled corticosteroids.

DETAILED DESCRIPTION:
This was a phase III, multicenter, randomized, double-blind active controlled 2-arm parallel group to compare superiority of CHF 1535 pressurised metered dose inhaler (pMDI) compared with CHF 718 pMDI, in subjects with asthma on medium or high dose inhaled corticosteroids, with regard to change from baseline in forced expiratory volume in the first second (FEV1) Area under the Curve Calculated Between Time 0 and 12 Hours (AUC0-12h) at Week 12.

After screening, eligible subjects entered a 2-week run-in period using CHF 718 (BDP) pMDI 100µg, followed by a 12-week double-blind, treatment period. Screened subjects who were on a medium dose inhaled corticosteroid (ICS) or medium dose ICS-long-acting β2-adrenergic receptor agonists (LABA) prior to the study, received CHF 718 pMDI 100µg 2 inhalations twice daily (BID) i.e. total daily dose (TDD) 400µg) during the 2-week run in period. Screened subjects who were on a high dose ICS prior to the study received CHF 718 pMDI 100µg 4 inhalations BID (TDD 800µg) during the 2-week run in period.

Following the run-in period, eligible subjects were randomized to one of two study drug arms (using a 1:1 allocation ratio) for 12 weeks. A total of 6 clinic visits (V), (V0-V5) and a follow-up call (V6) were performed during the study.

During the study, daily symptoms, rescue medication use, and compliance with the study drug were recorded via a subject-specific electronic diary (eDiary). Concomitant medications and adverse events (AEs) were assessed and recorded throughout the study. Vital signs measurements, physical exam, 12-lead electrocardiogram (ECG), peak expiratory flow (PEF), and spirometry measurements, including serial spirometry were performed and recorded. Symptoms were assessed using disease specific questionnaires. Routine hematology, blood chemistry, and urine pregnancy testing were performed before enrolment and at the end of study.

CHF 1535 pMDI = 200/6 μg pressurised metered dose inhaler (fixed combination of extrafine beclomethasone dipropionate [BDP] plus formoterol fumarate [FF]).

CHF 718 pMDI = 100 μg pressurised metered dose inhaler (extrafine beclomethasone dipropionate [BDP]).

ELIGIBILITY:
Inclusion Criteria (IC):

1. Informed consent: A signed and dated written informed consent obtained prior to any study-related procedures.
2. Sex and age: Male or female aged ≥18 and ≤75 years.
3. Diagnosis of asthma: A documented history of asthma for at least 1 year, with onset before age 40
4. Stable asthma therapy: Use of medium-dose ICS with or without a LABA or high-dose ICS alone for 3 months (at a stable dose for at least 4 weeks prior to screening).
5. Lung function: Subjects with a pre-bronchodilator FEV1 ≥40% and ≤85% of predicted, after appropriate washout from bronchodilators, at the screening and randomization visits. In addition, the absolute value of the first pre-dose FEV1 at randomization (V2) must be at least 80% of the pre-bronchodilator value attained at screening.
6. Reversibility post-bronchodilator: Subjects with a positive reversibility to bronchodilator at screening, defined as an increase in FEV1 > 12% and > 200mL compared to baseline within 30 minutes after 4 inhalations of albuterol hydrofluoroalkane (HFA) pMDI 90µg/actuation.

   Note for IC#5 and IC#6: In case the reversibility and/or quality threshold is not met at screening, the test can be performed once before randomization.
7. Female subjects:

   a. Women of childbearing potential (WOCBP) fulfilling one of the following criteria: i. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signing of the informed consent form and until the follow-up contact or ii. WOCBP with non-fertile male partners (contraception is not required in this case).

   b. Female subjects of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile as per definitions given in Appendix 2). Tubal ligation or partial surgical interventions are not acceptable. If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges).
8. Cooperative attitude and ability to demonstrate correct use of the pMDI inhalers and eDiary/peak flow meter.

Exclusion Criteria:

1. Pregnancy or lactation: where pregnancy is defined as the state of a female after conception and until termination of the gestation, confirmed by a positive pregnancy test (serum and urine pregnancy test to be performed at screening visit and urine pregnancy test to be performed prior to randomization).
2. Poor compliance with run-in medication or eDiary completion <50% before randomization.
3. History of "at risk" asthma: History of near-fatal asthma or of a past hospitalization for asthma in intensive care unit which, in the judgement of the investigator, may place the subject at undue risk.
4. Recent asthma exacerbation: Hospitalization, emergency room admission or use of systemic corticosteroids for an asthma exacerbation in the 4 weeks prior to screening visit or during the run-in period.
5. Unresolved respiratory tract infection (RTI) in the 4 weeks prior to the screening visit or during run-in period. Documented coronavirus disease 2019 (COVID-19) diagnosis within the last 8 weeks or complications from this disease, which have not resolved within 14 days prior to screening.
6. Unstable ICS dose during the 4 weeks prior to screening visit, including any change in dose, schedule, or formulation.
7. Use of systemic corticosteroid medication in the 4 weeks prior to screening or slow-release corticosteroids in the 12 weeks before screening.
8. Respiratory disorders other than asthma: History of a diagnosis of cystic fibrosis, bronchiectasis, Chronic Obstructive Pulmonary Disease (COPD), (as defined by the current Global Initiative for Chronic Obstructive Lung Disease [GOLD] Report), alpha-1 antitrypsin deficiency, or any other significant lung disease which may interfere with study evaluations.
9. Smoking status: Current smokers or ex-smokers with total cumulative exposure equal to or more than 10 pack-years or having stopped smoking within one year prior to screening visit.
10. E-cigarette status: Current e-cigarettes users at the time of the screening visit.
11. Cannabis usage: Current use of inhaled or oral cannabis products (e.g. marijuana).
12. Substance abuse: Subjects with a history of alcohol or substance/drug abuse within 12 months prior to screening.
13. Cardiovascular diseases: Subjects who have clinically significant cardiovascular condition such as, but not limited to, unstable ischemic heart disease, New York Heart Association (NYHA) Class III/IV heart failure, acute ischemic heart disease within one year prior to study entry, known history of atrial fibrillation or history of sustained and non-sustained cardiac arrhythmias diagnosed within the last 6 months prior to screening, not controlled with a rate control strategy. Note: Subjects with Permanent Atrial Fibrillation (for at least 6 months) with a resting ventricular rate <100/min, controlled with a rate control strategy (i.e., selective β-blocker, calcium channel blocker, pacemaker placement, digoxin, or ablation therapy) can be considered for the enrollment.
14. ECG criteria: An abnormal and clinically significant 12-lead electrocardiogram (ECG) which may impact the safety of the subject according to Investigator's judgement. In terms of the QTcF, subjects with QTcF >450ms for males or QTcF >470ms for females at screening or at randomization visits (criterion not applicable for subject with pacemaker or permanent atrial fibrillation).
15. Other medical conditions: Other active severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
16. Vaccination: Subjects having received a vaccination within 2 weeks prior to screening or during the run-in period.
17. Subjects' wellbeing: Subjects mentally or legally incapacitated, including but not limited to subjects who are institutionalized or incarcerated.
18. Hypersensitivity: Subjects with known intolerance, hypersensitivity or contraindication to treatment with ß2-agonists, ICS, or propellant gases/excipients.
19. Surgery: Subjects with major surgery in the 3 months prior to the screening visit or planned surgery during the study.
20. Additional treatment: Subjects treated with non-potassium sparing diuretics (unless administered as a fixed-dose combination with a potassium conserving drug or changed to potassium sparing before the screening), non-selective beta-blocking drugs, quinidine, quinidine-like anti-arrhythmic, or any medication with a QTc prolongation potential or a history of QTc prolongation.
21. Subjects treated with monoamine oxidase inhibitors (MAOIs) and tricyclic antidepressants.
22. Subjects with concomitant immunosuppressive therapy, use of oral or injected corticosteroids, anti-immunoglobulin E (IgE), anti-IL5 or other monoclonal or polyclonal antibodies within 12 weeks prior to screening.
23. Subjects who are receiving any therapy that could interfere with the study drugs according to investigator's opinion.
24. Participating in other investigational trial: Subjects who have received an investigational drug within 1 month or 5 half-lives (whichever is greater) prior to screening visit, or have been previously randomized in this trial, or are currently participating in another clinical trial.
25. Spacer: The need to use a spacer for correct self-administration of a pMDI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1377 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven F. Weinstein, M.D., Principal Investigator — Allergy and Asthma Specialists Medical Group and Research Center
Locations (91):
- United States (91):
  - Chiesi Clinical Trial Site 840858, Mobile, Alabama
  - Chiesi Clinical Trial Site 840895, Chandler, Arizona
  - Chiesi Clinical Trial Site 840856, Encinitas, California
  - Chiesi Clinical Trial Site 840843, Huntington Beach, California
  - Chiesi Clinical Trial Site 840860, Huntington Beach, California
  - Chiesi Clinical Trial Site 840896, Long Beach, California
  - Chiesi Clinical Trial Site 840883, Los Angeles, California
  - Chiesi Clinical Trial Site 840810, Los Angeles, California
  - Chiesi Clinical Trial Site 840869, Newport Beach, California
  - Chiesi Clinical Trial Site 840890, North Hollywood, California
  - Chiesi Clinical Trial Site 840808, Northridge, California
  - Chiesi Clinical Trial Site 840879, Pomona, California
  - Chiesi Clinical Trial Site 840868, Sacramento, California
  - Chiesi Clinical Trial Site 840849, San Diego, California
  - Chiesi Clinical Trial Site 840877, San Diego, California
  - Chiesi Clinical Trial Site 840861, San Jose, California
  - Chiesi Clinical Trial Site 840881, Westminster, California
  - Chiesi Clinical Trial Site 840873, Colorado Springs, Colorado
  - Chiesi Clinical Trial Site 840800, Denver, Colorado
  - Chiesi Clinical Trial Site 840820, Coral Gables, Florida
  - Chiesi Clinical Trial Site 840841, Cutler Bay, Florida
  - Chiesi Clinical Trial Site 840817, Greenacres City, Florida
  - Chiesi Clinical Trial Site 840822, Hialeah, Florida
  - Chiesi Clinical Trial Site 840838, Hialeah, Florida
  - Chiesi Clinical Trial Site 840864, Kissimmee, Florida
  - Chiesi Clinical Trial Site 840814, Miami, Florida
  - Chiesi Clinical Trial Site 840819, Miami, Florida
  - Chiesi Clinical Trial Site 840875, Miami, Florida
  - Chiesi Clinical Trial Site 840887, Miami, Florida
  - Chiesi Clinical Trial Site 840821, Miami, Florida
  - Chiesi Clinical Trial Site 840829, Miami, Florida
  - Chiesi Clinical Trial Site 840828, Miami, Florida
  - Chiesi Clinical Trial Site 840847, Miami, Florida
  - Chiesi Clinical Trial Site 840818, Miami, Florida
  - Chiesi Clinical Trial Site 840802, Miami, Florida
  - Chiesi Clinical Trial Site 840835, Miami, Florida
  - Chiesi Clinical Trial Site 840806, Miami, Florida
  - Chiesi Clinical Trial Site 840855, Miami, Florida
  - Chiesi Clinical Trial Site 840809, Miami Gardens, Florida
  - Chiesi Clinical Trial Site 840863, Miami Lakes, Florida
  - Chiesi Clinical Trial Site 840865, Miami Lakes, Florida
  - Chiesi Clinical Trial Site 840831, Miami Springs, Florida
  - Chiesi Clinical Trial Site 840839, Palmetto Bay, Florida
  - Chiesi Clinical Trial Site 840840, Pembroke Pines, Florida
  - Chiesi Clinical Trial Site 840827, Pembroke Pines, Florida
  - Chiesi Clinical Trial Site 840811, Port Saint Lucie, Florida
  - Chiesi Clinical Trial Site 840889, St. Petersburg, Florida
  - Chiesi Clinical Trial Site 840834, St. Petersburg, Florida
  - Chiesi Clinical Trial Site 840880, St. Petersburg, Florida
  - Chiesi Clinical Trial Site 840807, Tallahassee, Florida
  - Chiesi Clinical Trial Site 840871, Adairsville, Georgia
  - Chiesi Clinical Trial Site 840824, White Marsh, Maryland
  - Chiesi Clinical Trial Site 840826, North Dartmouth, Massachusetts
  - Chiesi Clinical Trial Site 840859, Columbia, Missouri
  - Chiesi Clinical Trial Site 840888, Saint Charles, Missouri
  - Chiesi Clinical Trial Site 840846, St Louis, Missouri
  - Chiesi Clinical Trial Site 840867, Bellevue, Nebraska
  - Chiesi Clinical Trial Site 840897, Henderson, Nevada
  - Chiesi Clinical Trial Site 840872, North Las Vegas, Nevada
  - Chiesi Clinical Trial Site 840836, Brick, New Jersey
  - Chiesi Clinical Trial Site 840851, Albuquerque, New Mexico
  - Chiesi Clinical Trial Site 840899, Monroe, North Carolina
  - Chiesi Clinical Trial Site 840852, Raleigh, North Carolina
  - Chiesi Clinical Trial Site 840866, Edmond, Oklahoma
  - Chiesi Clinical Trial Site 840878, Tulsa, Oklahoma
  - Chiesi Clinical Trial Site 840884, Grants Pass, Oregon
  - Chiesi Clinical Trial Site 840830, Medford, Oregon
  - Chiesi Clinical Trial Site 840853, Portland, Oregon
  - Chiesi Clinical Trial Site 840885, Warwick, Rhode Island
  - Chiesi Clinical Trial Site 840892, Anderson, South Carolina
  - Chiesi Clinical Trial Site 840844, Columbia, South Carolina
  - Chiesi Clinical Trial Site 840850, Greenville, South Carolina
  - Chiesi Clinical Trial Site 840894, Rock Hill, South Carolina
  - Chiesi Clinical Trial Site 840891, Spartanburg, South Carolina
  - Chiesi Clinical Trial Site 840812, Knoxville, Tennessee
  - Chiesi Clinical Trial Site 840815, Baytown, Texas
  - Chiesi Clinical Trial Site 840874, Boerne, Texas
  - Chiesi Clinical Trial Site 840845, Carrollton, Texas
  - Chiesi Clinical Trial Site 840876, Dallas, Texas
  - Chiesi Clinical Trial Site 840803, El Paso, Texas
  - Chiesi Clinical Trial Site 840833, Houston, Texas
  - Chiesi Clinical Trial Site 840862, McKinney, Texas
  - Chiesi Clinical Trial Site 840816, McKinney, Texas
  - Chiesi Clinical Trial Site 840842, San Antonio, Texas
  - Chiesi Clinical Trial Site 840857, San Antonio, Texas
  - Chiesi Clinical Trial Site 840823, San Antonio, Texas
  - Chiesi Clinical Trial Site 840801, Sugar Land, Texas
  - Chiesi Clinical Trial Site 840893, Murray, Utah
  - Chiesi Clinical Trial Site 840837, Riverton, Utah
  - Chiesi Clinical Trial Site 840882, Bellingham, Washington
  - Chiesi Clinical Trial Site 840870, Greenfield, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pelaia C, Crimi C, Vatrella A, Tinello C, Terracciano R, Pelaia G. Molecular Targets for Biological Therapies of Severe Asthma. Front Immunol. 2020 Nov 30;11:603312. doi: 10.3389/fimmu.2020.603312. eCollection 2020. PMID 33329598
- [Background] Roger JH, Bratton DJ, Mayer B, Abellan JJ, Keene ON. Treatment policy estimands for recurrent event data using data collected after cessation of randomised treatment. Pharm Stat. 2019 Jan;18(1):85-95. doi: 10.1002/pst.1910. Epub 2018 Nov 8. PMID 30406948
- [Background] Kardas G, Kuna P, Panek M. Biological Therapies of Severe Asthma and Their Possible Effects on Airway Remodeling. Front Immunol. 2020 Jun 18;11:1134. doi: 10.3389/fimmu.2020.01134. eCollection 2020. PMID 32625205
- [Background] Kippelen P, Anderson SD, Hallstrand TS. Mechanisms and Biomarkers of Exercise-Induced Bronchoconstriction. Immunol Allergy Clin North Am. 2018 May;38(2):165-182. doi: 10.1016/j.iac.2018.01.008. PMID 29631728
- [Background] Chau-Etchepare F, Hoerger JL, Kuhn BT, Zeki AA, Haczku A, Louie S, Kenyon NJ, Davis CE, Schivo M. Viruses and non-allergen environmental triggers in asthma. J Investig Med. 2019 Oct;67(7):1029-1041. doi: 10.1136/jim-2019-001000. Epub 2019 Jul 27. PMID 31352362
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Forno E, Celedon JC. Asthma and ethnic minorities: socioeconomic status and beyond. Curr Opin Allergy Clin Immunol. 2009 Apr;9(2):154-60. doi: 10.1097/aci.0b013e3283292207. PMID 19326508
- [Background] Zein JG, Udeh BL, Teague WG, Koroukian SM, Schlitz NK, Bleecker ER, Busse WB, Calhoun WJ, Castro M, Comhair SA, Fitzpatrick AM, Israel E, Wenzel SE, Holguin F, Gaston BM, Erzurum SC; Severe Asthma Research Program. Impact of Age and Sex on Outcomes and Hospital Cost of Acute Asthma in the United States, 2011-2012. PLoS One. 2016 Jun 13;11(6):e0157301. doi: 10.1371/journal.pone.0157301. eCollection 2016. PMID 27294365
- [Background] Global Initiative for Asthma (GINA): global strategy for asthma management and prevention. 2021 update. (2021). Available from: www.ginasthma.org.
- [Background] Davis J, Trudo F, Siddall J, Small M. Burden of asthma among patients adherent to ICS/LABA: A real-world study. J Asthma. 2019 Mar;56(3):332-340. doi: 10.1080/02770903.2018.1455858. Epub 2018 Apr 6. PMID 29624458
- [Background] Bateman ED, Boushey HA, Bousquet J, Busse WW, Clark TJ, Pauwels RA, Pedersen SE; GOAL Investigators Group. Can guideline-defined asthma control be achieved? The Gaining Optimal Asthma ControL study. Am J Respir Crit Care Med. 2004 Oct 15;170(8):836-44. doi: 10.1164/rccm.200401-033OC. Epub 2004 Jul 15. PMID 15256389
- [Background] Lee LK, Obi E, Paknis B, Kavati A, Chipps B. Asthma control and disease burden in patients with asthma and allergic comorbidities. J Asthma. 2018 Feb;55(2):208-219. doi: 10.1080/02770903.2017.1316394. Epub 2017 Jun 6. PMID 28586296
- [Background] Kerstjens HAM, Maspero J, Chapman KR, van Zyl-Smit RN, Hosoe M, Tanase AM, Lavecchia C, Pethe A, Shu X, D'Andrea P; IRIDIUM trial investigators. Once-daily, single-inhaler mometasone-indacaterol-glycopyrronium versus mometasone-indacaterol or twice-daily fluticasone-salmeterol in patients with inadequately controlled asthma (IRIDIUM): a randomised, double-blind, controlled phase 3 study. Lancet Respir Med. 2020 Oct;8(10):1000-1012. doi: 10.1016/S2213-2600(20)30190-9. Epub 2020 Jul 9. PMID 32653074
- [Background] Sobieraj DM, Baker WL, Nguyen E, Weeda ER, Coleman CI, White CM, Lazarus SC, Blake KV, Lang JE. Association of Inhaled Corticosteroids and Long-Acting Muscarinic Antagonists With Asthma Control in Patients With Uncontrolled, Persistent Asthma: A Systematic Review and Meta-analysis. JAMA. 2018 Apr 10;319(14):1473-1484. doi: 10.1001/jama.2018.2757. PMID 29554174
- [Background] Averell CM, Laliberte F, Duh MS, Wu JW, Germain G, Faison S. Characterizing Real-World Use Of Tiotropium In Asthma In The USA. J Asthma Allergy. 2019 Oct 7;12:309-321. doi: 10.2147/JAA.S216932. eCollection 2019. PMID 31632091
- [Background] Paggiaro P, Corradi M, Latorre M, Raptis H, Muraro A, Gessner C, Siergiejko Z, Scuri M, Petruzzelli S. High strength extrafine pMDI beclometasone/formoterol (200/6 mug) is effective in asthma patients not adequately controlled on medium-high dose of inhaled corticosteroids. BMC Pulm Med. 2016 Dec 9;16(1):180. doi: 10.1186/s12890-016-0335-9. PMID 27938358
- [Background] Papi A, Paggiaro PL, Nicolini G, Vignola AM, Fabbri LM; Inhaled Combination Asthma Treatment versus SYmbicort (ICAT SY) Study Group. Beclomethasone/formoterol versus budesonide/formoterol combination therapy in asthma. Eur Respir J. 2007 Apr;29(4):682-9. doi: 10.1183/09031936.00095906. Epub 2006 Nov 15. PMID 17107988
- [Background] Papi A, Paggiaro P, Nicolini G, Vignola AM, Fabbri LM; ICAT SE study group. Beclomethasone/formoterol vs fluticasone/salmeterol inhaled combination in moderate to severe asthma. Allergy. 2007 Oct;62(10):1182-8. doi: 10.1111/j.1398-9995.2007.01493.x. PMID 17845589
- [Background] Corradi M, Spinola M, Petruzzelli S, Kuna P. High-dose beclometasone dipropionate/formoterol fumarate in fixed-dose combination for the treatment of asthma. Ther Adv Respir Dis. 2016 Oct;10(5):492-502. doi: 10.1177/1753465816654442. Epub 2016 Jun 23. PMID 27340255
- [Background] Virchow JC, Kuna P, Paggiaro P, Papi A, Singh D, Corre S, Zuccaro F, Vele A, Kots M, Georges G, Petruzzelli S, Canonica GW. Single inhaler extrafine triple therapy in uncontrolled asthma (TRIMARAN and TRIGGER): two double-blind, parallel-group, randomised, controlled phase 3 trials. Lancet. 2019 Nov 9;394(10210):1737-1749. doi: 10.1016/S0140-6736(19)32215-9. Epub 2019 Sep 30. PMID 31582314
- [Background] Lee LA, Bailes Z, Barnes N, Boulet LP, Edwards D, Fowler A, Hanania NA, Kerstjens HAM, Kerwin E, Nathan R, Oppenheimer J, Papi A, Pascoe S, Brusselle G, Peachey G, Sule N, Tabberer M, Pavord ID. Efficacy and safety of once-daily single-inhaler triple therapy (FF/UMEC/VI) versus FF/VI in patients with inadequately controlled asthma (CAPTAIN): a double-blind, randomised, phase 3A trial. Lancet Respir Med. 2021 Jan;9(1):69-84. doi: 10.1016/S2213-2600(20)30389-1. Epub 2020 Sep 9. PMID 32918892
- [Background] Fink JB, Colice GL, Hodder R. Inhaler devices for patients with COPD. COPD. 2013 Aug;10(4):523-35. doi: 10.3109/15412555.2012.761960. Epub 2013 Mar 28. PMID 23537191
- [Background] Lipworth B, Manoharan A, Anderson W. Unlocking the quiet zone: the small airway asthma phenotype. Lancet Respir Med. 2014 Jun;2(6):497-506. doi: 10.1016/S2213-2600(14)70103-1. PMID 24899370
- [Background] Juniper EF, Bousquet J, Abetz L, Bateman ED; GOAL Committee. Identifying 'well-controlled' and 'not well-controlled' asthma using the Asthma Control Questionnaire. Respir Med. 2006 Apr;100(4):616-21. doi: 10.1016/j.rmed.2005.08.012. Epub 2005 Oct 13. PMID 16226443
- [Background] Juniper EF, O'Byrne PM, Guyatt GH, Ferrie PJ, King DR. Development and validation of a questionnaire to measure asthma control. Eur Respir J. 1999 Oct;14(4):902-7. doi: 10.1034/j.1399-3003.1999.14d29.x. PMID 10573240
- [Background] Roland NJ, Bhalla RK, Earis J. The local side effects of inhaled corticosteroids: current understanding and review of the literature. Chest. 2004 Jul;126(1):213-9. doi: 10.1378/chest.126.1.213. PMID 15249465
- [Background] Ellepola AN, Samaranayake LP. Inhalational and topical steroids, and oral candidosis: a mini review. Oral Dis. 2001 Jul;7(4):211-6. PMID 11575870
- [Background] Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, Casale TB, Chanez P, Enright PL, Gibson PG, de Jongste JC, Kerstjens HA, Lazarus SC, Levy ML, O'Byrne PM, Partridge MR, Pavord ID, Sears MR, Sterk PJ, Stoloff SW, Sullivan SD, Szefler SJ, Thomas MD, Wenzel SE; American Thoracic Society/European Respiratory Society Task Force on Asthma Control and Exacerbations. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med. 2009 Jul 1;180(1):59-99. doi: 10.1164/rccm.200801-060ST. PMID 19535666
- [Background] Virchow JC, Backer V, de Blay F, Kuna P, Ljorring C, Prieto JL, Villesen HH. Defining moderate asthma exacerbations in clinical trials based on ATS/ERS joint statement. Respir Med. 2015 May;109(5):547-56. doi: 10.1016/j.rmed.2015.01.012. Epub 2015 Feb 3. PMID 25676887
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Background] Fagerland MW, Lydersen S, Laake P. Recommended confidence intervals for two independent binomial proportions. Stat Methods Med Res. 2015 Apr;24(2):224-54. doi: 10.1177/0962280211415469. Epub 2011 Oct 13. PMID 21996567
- [Derived] Weinstein S, Legramandi L, Mathews KS, Passineau H, Seregni L, Gandini G, Cretarola L, Foti M, Skloot G, Hernandez G. Improved lung function with beclomethasone/formoterol versus beclomethasone alone in asthma: the FORCE2 study. J Asthma. 2025 Nov 22:1-7. doi: 10.1080/02770903.2025.2589794. Online ahead of print. PMID 41231513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, 1377 participants were enrolled into the study; of these, 576 met eligibility criteria and were randomized to treatment.
Groups:
- CHF 1535 pMDI: CHF 1535 pMDI 800/24µg TDD
  Beclomethasone Dipropionate/Formoterol Fumarate: pressurized inhalation solution BDP/FF 200/6 µg
- CHF 718 pMDI: CHF 718 pMDI 800µg TDD
  Beclomethasone Dipropionate: pressurized inhalation solution BDP 100 µg
Period: Overall Study
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Started | 287 | 289
Completed | 276 | 267
Not Completed | 11 | 22
Not completed — Withdrawal by Subject | 3 | 10
Not completed — Randomization error | 3 | 7
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Patient refused treatment | 1 | 0
Not completed — Patient could not travel to the study site | 1 | 0
Not completed — Technical issues with the masterscope | 0 | 3
Not completed — Patient moved to a different state | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI | Total
Number analyzed (Participants) | 283 | 280 | 563
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 231 | 237 | 468
  >=65 years | 52 | 43 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (14.1) | 50.3 (14.1) | 50.9 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 202 | 412
  Male | 73 | 78 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 154 | 165 | 319
  Not Hispanic or Latino | 129 | 113 | 242
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 6 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 59 | 49 | 108
  White | 216 | 220 | 436
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 283 | 280 | 563
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.90 (6.93) | 30.86 (7.27) | 30.88 (7.09)
Time since first asthma diagnosis [Mean (Standard Deviation); unit: months] | 474.6 (173.6) | 468.4 (180.9) | 471.5 (177.1)
Asthma medication at study entry [Count of Participants; unit: Participants] — ICS=Inhaled Corticosteroid LABA=Long-acting β2-adrenergic Receptor Agonists
  Participants
    Inhaled Corticosteroid/Long-acting β2-adrenergic Receptor Agonists (ICS/LABA) combination | 234 | 230 | 464
    ICS/LABA fixed combination | 228 | 221 | 449
    ICS+LABA free combination | 6 | 9 | 15
    High-dose ICS | 3 | 5 | 8
    Medium-dose ICS | 46 | 45 | 91
Number of asthma exacerbations in the 4 weeks prior to screening [Count of Participants; unit: Participants]
  0 | 283 | 280 | 563
  1+ | 0 | 0 | 0
Time since last documented exacerbation [Mean (Standard Deviation); unit: months] — Population: Data presented are for the number of subjects with available data.
  months
    number analyzed (Participants) | 43 | 53 | 96
    (all) | 52.4 (85.4) | 43.3 (87.9) | 47.3 (86.5)
Treatment of the most recent exacerbation [Count of Participants; unit: Participants] — Population: Data presented are for the number of subjects with available data.
  Participants
    Systemic corticosteroids: number analyzed (Participants) | 37 | 45 | 82
    Systemic corticosteroids | 35 | 43 | 78
    Hospitalisation: number analyzed (Participants) | 37 | 45 | 82
    Hospitalisation | 1 | 0 | 1
    Emergency room: number analyzed (Participants) | 37 | 45 | 82
    Emergency room | 12 | 7 | 19
Smoking status at screening [Count of Participants; unit: Participants]
  Non-smoker | 250 | 244 | 494
  Ex-smoker | 33 | 36 | 69
  Current smoker | 0 | 0 | 0
Smoking duration [Mean (Standard Deviation); unit: years] — Population: Data available only for ex-smokers.
  years
    number analyzed (Participants) | 33 | 36 | 69
    (all) | 13.58 (10.00) | 12.67 (9.29) | 13.11 (9.57)
Number of pack-years [Mean (Standard Deviation); unit: pack-years] — Pack-year: is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. Population: Data available only for ex-smokers.
  pack-years
    number analyzed (Participants) | 33 | 36 | 69
    (all) | 2.9 (2.7) | 3.7 (3.1) | 3.3 (2.9)
Electronic cigarettes - Smoking status at screening [Count of Participants; unit: Participants]
  Non-smoker | 283 | 280 | 563
  Ex-smoker | 0 | 0 | 0
  Current smoker | 0 | 0 | 0
FEV1 -- At baseline [Mean (Standard Deviation); unit: liters] — Forced Expiratory Volume in the First Second (FEV1).
  The baseline value was the arithmetic mean of the pre-dose FEV1 measurements (45 minutes and 15 minutes pre-dose) collected at Week 0 (V2). If one of the two pre-dose values was missing, the baseline was equal to the available pre-dose value. Otherwise, in case of both pre-dose measurements missing the baseline value was considered as missing. Population: Data presented are for the number of subjects with available data.
  liters
    number analyzed (Participants) | 283 | 279 | 562
    (all) | 1.850 (0.535) | 1.860 (0.559) | 1.855 (0.546)
FEV1 (% of predicted normal value) at baseline [Mean (Standard Deviation); unit: percent of predicted] — FEV1=Forced expiratory volume in the first second Population: Data presented are for the number of subjects with available data.
  percent of predicted
    number analyzed (Participants) | 283 | 279 | 562
    (all) | 64.104 (10.651) | 63.033 (10.739) | 63.572 (10.698)
FVC at baseline [Mean (Standard Deviation); unit: liters] — Forced Vital Capacity (FVC)
  liters | 2.661 (0.899) | 2.614 (0.945) | 2.637 (0.922)
ACQ score at baseline [Mean (Standard Deviation); unit: score] — ACQ=Asthma Control Questionnaire©
  ACQ-7:
  Assess asthma symptoms over last 7 days (night-time awakenings due to symptoms, morning symptoms, activity limitation, shortness of breath, wheezing), average daily rescue medication use, and current FEV1 percent predicted. Score scale: 0=totally controlled; 6=severely uncontrolled.
  ACQ-5:
  Assess asthma symptoms over last 7 days, consists of 5 items derived from the first 5 questions of ACQ7. Score scale: 0=totally controlled; 6=severely uncontrolled. Population: Data presented are for the number of subjects with available data.
  ACQ=Asthma Control Questionnaire©
  score
    ACQ-7: number analyzed (Participants) | 278 | 276 | 554
    ACQ-7 | 1.30 (0.88) | 1.25 (0.87) | 1.28 (0.88)
    ACQ-5 | 0.92 (0.95) | 0.88 (0.98) | 0.90 (0.96)

OUTCOME MEASURES:

1. Primary Outcome: 1_Change From Baseline in FEV1 AUC0-12h Normalised by Time at Week 12
Description: The pre-dose FEV1 at baseline (i.e. pre-dose on Week 0 [Visit 2]) and the FEV1 AUC0-12h normalised by time at Week 12 (Visit 5) are presented by treatment group in the ITT population, as change from baseline.
  AUC0=12h Area under the curve calculated between time 0 and 12 hours
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: Intention-to-treat (ITT) population: all randomised subjects who received at least one administration of the study drug.
  Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group).
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 272 | 258
liter | 0.279 [0.248 to 0.309] | 0.174 [0.143 to 0.206]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Change from baseline Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = 0.104, 95% CI 2-sided [0.061 to 0.148]

2. Secondary Outcome: 2_Change From Baseline in Peak FEV1 Within the First 3 Hours Post-dose at Week 12
Description: The peak FEV1 at baseline (i.e. pre-dose on Week 0 [V2]) and the peak FEV1 within the first 3 hours post-dose at Week 12 (V5) are presented by treatment group in the ITT population, as change from baseline.
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 276 | 264
liter | 0.419 [0.385 to 0.453] | 0.295 [0.260 to 0.330]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = 0.124, 95% CI 2-sided [0.076 to 0.173]

3. Secondary Outcome: 3_Change From Baseline in FEV1 AUC0-12h Normalised by Time at Week 0
Description: The pre-dose FEV1 at baseline (i.e. pre-dose on Week 0 [V2]) and the FEV1 AUC0-12h normalised by time at Week 0 (V2, post-dose) are presented by treatment group in the ITT population, as change from baseline.
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 278 | 277
liter | 0.250 [0.223 to 0.276] | 0.149 [0.122 to 0.175]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = 0.101, 95% CI 2-sided [0.063 to 0.139]

4. Secondary Outcome: 4_Change From Baseline in Peak FEV1 Within the First 3 Hours Post-dose at Week 0
Description: The peak FEV1 at baseline (i.e. pre-dose on Week 0 [V2]) and the peak FEV1 within the first 3 hours post-dose at Week 0 (V2, post-dose) are presented by treatment group in the ITT population, as change from baseline.
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and 3 h post dose on Week 0.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 278 | 277
liter | 0.374 [0.345 to 0.404] | 0.262 [0.233 to 0.291]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, ANCOVA; Adjusted mean difference = 0.113, 95% CI 2-sided [0.071 to 0.154]

5. Secondary Outcome: 5_Change From Baseline in Trough FEV1 at Week 12
Description: The trough FEV1 at baseline (i.e. pre-dose on Week 0 [V2]), the trough FEV1 at Week 12 (V5) and the change from baseline in trough FEV1 at Week 12 (V5) are presented by treatment group in the ITT population, as change from baseline.
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 274 | 264
liter | 0.212 [0.179 to 0.244] | 0.143 [0.110 to 0.176]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, ANCOVA; Adjusted mean difference = 0.069, 95% CI 2-sided [0.023 to 0.115]

6. Secondary Outcome: 6_Change From Baseline in Pre-dose Morning FEV1 at Weeks 4, 8 and 12
Description: The pre-dose MORNING FEV1 at baseline (i.e. pre-dose on Week 0 [V2]) and the pre-dose morning FEV1 at Week 4 (V3), Week 8 (V4) and Week 12 (V5) are presented by treatment group in the ITT population, as change from baseline.
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and Week 4, Week 8, Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 283 | 280
liter
  Week 4 (V3): number analyzed (Participants) | 280 | 272
  Week 4 (V3) | 0.152 [0.121 to 0.182] | 0.107 [0.076 to 0.139]
  Week 8 (V4): number analyzed (Participants) | 279 | 270
  Week 8 (V4) | 0.188 [0.154 to 0.222] | 0.147 [0.113 to 0.182]
  Week 12 (V5): number analyzed (Participants) | 278 | 267
  Week 12 (V5) | 0.162 [0.132 to 0.193] | 0.120 [0.088 to 0.151]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Change from baseline -- Week 4 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.050, ANCOVA; Adjusted mean difference = 0.044, 95% CI 2-sided [0.000 to 0.088]
Statistical Analysis 2: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 2_Change from baseline -- Week 8 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.098, ANCOVA; Adjusted mean difference = 0.041, 95% CI 2-sided [-0.007 to 0.089]
Statistical Analysis 3: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 3_Change from baseline -- Week 12 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.056, ANCOVA; Adjusted mean difference = 0.043, 95% CI 2-sided [-0.001 to 0.086]

7. Secondary Outcome: 7_Proportion of Pre-dose Morning FEV1 Responders at Weeks 4, 8 and 12
Description: The proportion of pre-dose MORNING FEV1 responders at Week 4 (V3), Week 8 (V4) and Week 12 (V5) are presented by treatment group in the ITT population. The proportion of subjects classified as pre-dose morning FEV1 responders (i.e. those subjects who had change from baseline in pre-dose morning FEV1 ≥100 mL).
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and Week 4, Week 8, Week 12.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 283 | 280
Participants
  Week 4 (V3) | 154 | 130
  Week 8 (V4) | 162 | 141
  Week 12 (V5) | 162 | 125
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Responders at Week 4; Test type: Superiority; p = 0.098, Logistic regression model; Odds Ratio (OR) = 1.327, 95% CI 2-sided [0.949 to 1.855]
Statistical Analysis 2: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 2_Responders at Week 8; Test type: Superiority; p = 0.180, Logistic regression model; Odds Ratio (OR) = 1.262, 95% CI 2-sided [0.898 to 1.772]
Statistical Analysis 3: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 3_Responders at Week 12; Test type: Superiority; p = 0.009, Logistic regression model; Odds Ratio (OR) = 1.568, 95% CI 2-sided [1.117 to 2.203]

8. Secondary Outcome: 8_Proportion of Trough FEV1 Responders at Week 12
Description: The proportion of trough FEV1 responders at Week 12 (V5) are presented by treatment group in the ITT population.
  The proportion of subjects classified as trough FEV1 responders (i.e. those subjects who had change from baseline in trough FEV1 ≥100 mL).
  FEV1=Forced Expiratory Volume in the First Second
Time Frame: Baseline (pre-dose on Week 0) and Week 4, Week 8, Week 12.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 283 | 280
Participants | 181 | 136
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Responders at Week 12; Test type: Superiority; p < 0.001, Logistic regression model; Odds Ratio (OR) = 1.822, 95% CI 2-sided [1.284 to 2.587]

9. Secondary Outcome: 9_Change From Baseline in Average Morning Peak Expiratory Flow (PEF) Over the 12-Week Treatment Period
Description: The average MORNING PEF at baseline (i.e. average morning "Best PEF" values during the run-in period, over each inter-visit period and over the 12-week treatment period are presented by treatment group in the ITT population), as change from baseline.
  PEF=Peak Expiratory Flow
Time Frame: Baseline (Week 0) to Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter/min
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 279 | 277
liter/min | 13.45 [9.58 to 17.32] | 4.67 [0.77 to 8.56]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Change From Baseline; Week 0 -- Week 12 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.002, ANCOVA; Adjusted mean difference = 8.78, 95% CI 2-sided [3.30 to 14.27]

10. Secondary Outcome: 10_Change From Baseline in Average Evening Peak Expiratory Flow (PEF) Over the 12-Week Treatment Period
Description: The average EVENING PEF at baseline (i.e. average evening "Best PEF" values during the run-in period, see Section 9.7.1.4), over each inter-visit period and over the 12-week treatment period are presented by treatment group in the ITT population, as change from baseline.
  PEF=Peak Expiratory Flow
Time Frame: Baseline (Week 0) to Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: liter/min
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 280 | 277
liter/min | 10.27 [6.46 to 14.08] | 1.54 [-2.31 to 5.38]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.002, ANCOVA; Adjusted mean difference = 8.73, 95% CI 2-sided [3.32 to 14.14]

11. Secondary Outcome: 11_Change From Baseline in ACQ-7 Score and ACQ-5 Score at Week 12
Description: The ACQ-7 and ACQ-5 scores at baseline (i.e. pre-dose on Week 0 [V2]) and at Week 12 (V5) are presented by treatment group in the ITT population, as change from baseline; only patients who provided required data at baseline and at specified times are included in the calculation.
  Asthma control was evaluated during the treatment period (Week 0 to Week 12 [V2-V5])/end of treatment (ET) if applicable, using ACQ-7; first 6 items refer to symptoms and rescue use in the previous 7 days. The 7th item, filled in by the clinical staff, was the FEV1 (% predicted) recorded at 15 min pre-dose, measured at each visit during the treatment period. ACQ-5 has 5 items on adequacy of asthma control.
  ACQ-7:
  Assess asthma symptoms over last 7 days (night-time awakenings due to symptoms, morning symptoms, activity limitation, shortness of breath, wheezing), average daily rescue medication use, and current FEV1 percent predicted. Score scale: 0=totally controlled; 6=severely uncontrolled.
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 283 | 280
score
  ACQ-7: number analyzed (Participants) | 272 | 260
  ACQ-7 | -0.414 [-0.484 to -0.345] | -0.302 [-0.373 to -0.231]
  ACQ-5: number analyzed (Participants) | 279 | 269
  ACQ-5 | -0.413 [-0.481 to -0.345] | -0.433 [-0.503 to -0.364]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 1_Change From Baseline in ACQ-7 at Week 12 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.026, ANCOVA; Adjusted mean difference = -0.112, 95% CI 2-sided [-0.211 to -0.013]
Statistical Analysis 2: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; 2_Change from baseline in ACQ-5 at Week 12 Statistical analysis used all available data and imputed missing data (i.e., whether due to missed visits, unperformed or unevaluable assessments at intermediate timepoints, or early study discontinuation) in ITT population (overall population N=283 in CHF 1535 pMDI 800/24 μg study group; N=280 in the CHF 718 pMDI 800 μg study group); Test type: Superiority; p = 0.686, ANCOVA; Adjusted mean difference = 0.020, 95% CI 2-sided [-0.077 to 0.118]

12. Secondary Outcome: 12_Change From Baseline in Percentage of Rescue Medication-free Days Over the 12-Week Treatment Period
Description: The percentage of rescue medication-free days at baseline (i.e. percentage of days during the run-in period with no rescue medication), over each inter-visit period and over the 12-week treatment period are presented by treatment group in the ITT population, as change from baseline.
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 282 | 279
percentage of days | 17.923 [15.457 to 20.388] | 14.103 [11.617 to 16.589]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.033, ANCOVA; Adjusted mean difference = 3.820, 95% CI 2-sided [0.310 to 7.330]

13. Secondary Outcome: 13_Change From Baseline in Percentage of Asthma Symptom-free Days Over the 12-Week Treatment Period
Description: The percentage of asthma symptom-free days at baseline (i.e. percentage of days during the run-in period with no asthma symptom, over each inter-visit period and over the 12-week treatment period are presented by treatment group in the ITT population, as change from baseline.
Time Frame: Baseline (pre-dose on Week 0) and Week 12.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
Number analyzed (Participants) | 223 | 212
percentage of days | 20.872 [17.908 to 23.836] | 17.092 [14.098 to 20.086]
Statistical Analysis 1: Comparison: CHF 1535 pMDI vs CHF 718 pMDI; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.078, ANCOVA; Adjusted mean difference = 3.780, 95% CI 2-sided [-0.425 to 7.985]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were reported from the time of patient informed consent signature until study completion at week 12 or at study discontinuation.
Description: Treatment-emergent AEs (TEAEs) were defined as AEs with date of first randomised study treatment intake as AE onset date or the date of study completion/discontinuation.
  Safety population: all randomised subjects who received at least one administration of the study drug.
Arm/Group | CHF 1535 pMDI | CHF 718 pMDI
All-Cause Mortality (participants affected / at risk) | 0/283 | 0/280
Serious Adverse Events (participants affected / at risk) | 3/283 | 0/280
Other Adverse Events (participants affected / at risk) | 44/283 | 53/280
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 1535 pMDI (N=283) | CHF 718 pMDI (N=280)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 1535 pMDI (N=283) | CHF 718 pMDI (N=280)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Bronchitis (Infections and infestations) | 0 (0) | 3 (3)
COVID-19 (Infections and infestations) | 4 (4) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (8) | 7 (7)
Oral candidiasis (Infections and infestations) | 3 (3) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 14 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (2)
Hypertension (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this study may be published or presented at scientific meetings. If a publication is presented by the Investigator, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor to Chiesi before submission.

DOCUMENTS (2):
  • Study Protocol (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT05292586/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT05292586/SAP_001.pdf